CLINICAL TRIAL: NCT01803035
Title: A Phase II, Randomised, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Two Doses of LTX-109 (1 % and 2 %) Versus Placebo in Impetigo
Brief Title: A Phase II Study to Evaluate the Efficacy and Safety of Two Doses of LTX-109 in Impetigo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lytix Biopharma AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C12-109-04
Record Dates: First submitted 2013-02-21; First posted 2013-03-04 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Non-bullous Impetigo
Keywords: Impetigo; LTX-109; Topical; Antibiotic; Placebo; Lytic; Peptide; Gram Positive
MeSH Terms: conditions — Impetigo

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 % LTX-109 (Experimental): LTX-109 topical gel in 1 % strength
  Interventions: Drug: LTX-109 1 %
- 2 % LTX-109 (Experimental): LTX-109 topical gel in 2 % strength
  Interventions: Drug: LTX-109 2 %
- Placebo (Placebo Comparator): Placebo gel, containing all ingredients except LTX-109
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: LTX-109 1 %
  Arms: 1 % LTX-109
Drug: LTX-109 2 %
  Arms: 2 % LTX-109
Drug: Placebo gel
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy of the topical antibiotic LTX-109 in terms of clinical and microbiological response in treatment of impetigo.

DETAILED DESCRIPTION:
The study will be a randomized, double-blind, placebo controlled study. Up to 210 patients will be enrolled to three treatment groups who will receive 1 % LTX-109, 2 % LTX-109 or placebo three times daily (TID) for 5 days. Patients will be randomized to receive LTX-109 or placebo at a ratio of 1:1 at each of the doses.

Patients ≥2 years with non-bullous impetigo will be enrolled in the study. Study candidacy will be determined by a dermatological examination, medical history, clinical diagnosis of non-bullous impetigo and a positive Gram-stain. Patients meeting eligibility will be randomized to one of the treatment groups.

A safety visit will be performed at Day 4. Clinical response will be evaluated by clinical success, clinical improvement or clinical failure according to definitions in the protocol at one or more of the visits - Day 4 (-1), Day 6 (+2) and Day 12 (+2), and will be derived from the Skin Infection Rating Scale (SIRS) score of the target lesion.

Bacteriological response will be evaluated by culture of swabs collected from the target lesion. Success or failure will be defined by presence or non-presence of the causative pathogen (bacteria isolated at baseline considered being the causative pathogen: S. aureus or S. pyogenes). Bacteriological swabs will be collected if pus/exudate is available at Day 4 (-1), Day 6 (+2) and Day 12 (+2), if there is exudate/pus available from the target lesion. No pus/exudate will be considered as elimination of the causative pathogen, and will be considered as bacteriological success.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 2 years of age.
* Signed written informed consent document by patient, parent, legal guardian or caretaker.
* Positive Gram-stain of target lesion showing Gram-positive cocci.
* Clinical diagnosis of primary non-bullous impetigo as per protocol.
* Candidate for treatment with topical antibacterial and have a Skin Infection Rating Scale (SIRS) of ≥ 4 with at least three of the five primary signs and symptoms present at baseline including a score of 1 or greater for exudate/pus.
* Total lesion area ≤ 20 cm2. Single lesion not to exceed 2 cm2.
* No known medical conditions that in the investigators opinion may interfere with study participation or put the patient at additional risk.

Exclusion Criteria:

* Unwillingness or inability of patient, parent, legal guardian or caretaker to comply with the requirements of the protocol.
* Presence of other skin disease at or near the investigational target area to be treated.
* The disease is so widespread or severe that, in the opinion of the investigator, the patient needs oral antibiotic treatment.
* History of hepatitis B or C, HIV, AIDS, or other immunodeficiency disease.
* Concurrent or recent scabies infection.
* Signs and symptoms of a current infection requiring antibiotic treatment.
* Tympanic temperature at Baseline > 38 °C (100.4 °F) in a pediatric patient or 37.8 °C (100 °F) in an adult patient.
* Use of systemic or topical antibiotics or steroids within 72 hours prior to study entry.
* Participation in any other clinical study or use of any other investigational drugs or investigational device within 30 days prior to treatment.
* Known allergy to any constituent of the study medication.
* Presence of secondarily-infected animal/human/insect bite or infected burn wound.
* Other reason which based on the discretion of the investigator makes the patient unsuitable for enrolment.
* Lactating or pregnant.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of LTX-109. | One year
  Efficacy of two doses 1% and 2% LTX-109 versus placebo will be measured by clinical response.
  Clinical response is defined as "Clinical success", "Clinical improvement" and "Clinical failure". Evaluation of the target lesion will be done at day 4, day 6 and day 12 and will be derived from Skin Infection Rating Scale (SIRS).

SECONDARY OUTCOMES:
Safety of topical administration in treatment of impetigo. | One year
  Safety will be monitored through physical examination, compliance with assigned treatment, and recording of adverse events occurring during the study period. Changes in clinical signs and symptoms will be recorded in the SIRS score. An assessment will be done of the target lesion and one overall assessment of the subject non-target lesions. A targeted physical examination will be done if any abnormalities occur.
  For the study analysis the number of patients with adverse events and the nature of the adverse events will be listed per treatment group.
Microbiological response of two doses of LTX-109 (1% and 2%) versus placebo in the treatment of impetigo. | One year
  Microbiological response will be measured by "Bacteriological Success" or "Bacteriological failure". The response will be derived from bacterial swab cultures, and presence or non-presence of the causative pathogen at each of the follow up visits, day 4, day 6, and day 12.

CONTACTS AND LOCATIONS:
Overall Officials: Daisy M Blanco, MD, Principal Investigator — Institute of Dermatology and Skin Surgery, Dr. Hubert Bogaert Diaz, Santo Domingo; Josefina Fernandez, MD, Principal Investigator — Dr. Robert Reid Cabral Children hospital, Santo Domingo
Locations (2):
- Dominican Republic (2):
  - Dr. Robert Reid Cabral Children Hospital, Santo Domingo
  - Institute of Dermatology and and Skin Surgery Dr. Hubert Bogaert Diaz, Santo Domingo